CLINICAL TRIAL: NCT03493802
Title: Assessment of Longitudinal Changes in Endothelial Function and Oxidative Stress in Normotensive Patients With Autosomal Dominant Polycystic Kidney Disease (ADPKD) - A Pilot Study
Brief Title: Assessment of Longitudinal Changes in Endothelial Function and Oxidative Stress in Normotensive Patients With ADPKD
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Maria V. Irazabal Mira, Principal Investigator, Mayo Clinic
Other Study IDs: 17-005944
Record Dates: First submitted 2018-03-23; First posted 2018-04-11 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: ADPKD; Endothelial dysfunction; Oxidative stress; NADPH oxidase 4 (NOX4); Mitochondria
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with a previous diagnosis of ADPKD: Patients that have been diagnosed with ADPKD and meet the study's inclusion criteria
- Healthy individuals as controls: Age and gender-matched healthy controls

SUMMARY:
The purpose of this study is to determine whether patients with autosomal dominant polycystic kidney disease (ADPKD) present with abnormal endothelial function, increased levels of NOX4 activity and mitochondrial abnormalities, contributing to oxidative stress from early stages that correlate with disease severity.

DETAILED DESCRIPTION:
Autosomal dominant polycystic kidney disease (ADPKD) is the most common monogenic and the fourth cause of end-stage renal disease (ESRD) in adults worldwide. Cardiovascular diseases are the most important non-cystic complications and continue to be the leading cause of premature mortality in these patients. Hypertension (HTN) is present in approximately 50% of the patients at early stages, and increases to nearly 100% at ESRD. Furthermore, HTN contributes to the underlying renal disease progression. Nitric oxide (NO) associated endothelium-dependent vasorelaxation has been shown to be impaired in small subcutaneous resistance vessels from patients with ADPKD before the development of HTN. However, the principal contributors to vascular dysfunction remain unclear.

The investigators broad objective is to evaluate the presence and extent of endothelial dysfunction and its association with oxidative stress in young normotensive patients with ADPKD, with the long term goal of timely intervention to slow the progression of the disease in these patients.

Participants in this study will have their endothelial function assessed using a non-invasive technique, peripheral arterial tonometry (PAT), which has been shown to be a useful, highly reproducible, and non-operator dependent method for non-invasive assessment of vascular health. The investigators will assess longitudinal changes in endothelial function using PAT with the intention of establishing if this methodology offers the potential of non-invasive measures of early vascular disease in young normotensive patients with ADPKD. Biochemical markers of endothelial dysfunction will be assessed concomitantly. In addition, the investigators will assess oxidative stress levels in these patients, with the intention of determining the association with endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

ADPKD Patients:

* ADPKD (based on Ravine et al. criteria)
* Class 1 B-D according to our imaging classification
* Male and female subjects 18 - 40 years of age, inclusive
* Estimated GFR> 60 mL/min/m2 (CKD-Epi equation)
* Systolic BP≤130mmHg without taking HTN medications
* Ability to provide written, informed consent

Healthy controls:

* Male and female subjects 18 - 40 years of age, inclusive
* estimated GFR> 60 mL/min/m2 (CKD-EPI equation)
* Systolic BP≤130mmHg without taking HTN medications
* Ability to provide written, informed consent

Exclusion Criteria:

ADPKD Patients:

* Class 2 according to our imaging classification
* Concomitant systemic disease in the kidney (e.g. lupus, hepatitis B or C, amyloidosis)
* Diabetes mellitus (fasting glucose > 126 mg/dL or treatment with insulin or oral hypoglycemics).
* Predicted urine protein excretion in urinalysis >1 g/24 hrs
* Abnormal urinalysis suggestive of concomitant glomerular disease
* Subjects having contraindications to, or interference with MRI assessments. [For example: ferromagnetic metal prostheses, aneurysm clips, severe claustrophobia, large abdominal/back tattoos, etc].
* Female subjects that are pregnant

Healthy controls:

* Previous personal or family history of kidney disease
* Concomitant systemic disease in the kidney (e.g. lupus, hepatitis B or C, amyloidosis)
* Diabetes mellitus (fasting glucose > 126 mg/dL or treatment with insulin or oral hypoglycemics).
* Presence of proteinuria
* Abnormal urinalysis suggestive glomerular disease
* Subjects having contraindications to, or interference with MRI assessments. [For example: ferromagnetic metal prostheses, aneurysm clips, severe claustrophobia, large abdominal/back tattoos, etc]
* Female subjects that are pregnant

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male and female patients with a previous diagnosis of ADPKD that meet the inclusion criteria. In addition, patients will be matched 2:1 to age and gender healthy controls. Exclusion criteria are listed in for ADPKD patients and healthy controls.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Assessment of endothelial function by Peripheral Artery Tonometry (PAT) | 18 months
  PAT is a novel non-invasive technology which records volume changes in the microcirculation of the digits in response to hyperemia, to measure peripheral vasodilator response as a measure for endothelial dysfunction.
NADPH oxidase 4 (NOX4) expression/activity | 18 months
  Determined by ELISA from plasma and urine
Mitochondrial DNA copy number | 18 months
  Plasma and urine levels of the mitochondria encoded genes cytochrome-c oxidase-3 (COX3) and nicotinamide adenine dinucleotide (NADH) dehydrogenase subunit-1 (ND1) determined by quantitative real-time polymerase chain reaction
Total kidney volume (TKV) | 18 months
  Determined by MRI
Renal blood flow (RBF) | 18 months
  Determined by MRI
Glomerular filtration rate (GFR) | 18 months
  Determination of iothalamate clearance

CONTACTS AND LOCATIONS:
Overall Officials: Maria V Irazabal, M.D., Ph.D., Principal Investigator — Mayo Translational PKD Center, Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials